CLINICAL TRIAL: NCT04841460
Title: Impact of Beef's Unique Food Matrix on Human Health - Cholesterol Metabolism and Voluntary Nutrient Intake in Men Consuming Low-fat and High-fat Ground Beef
Brief Title: Impact of Beef's Unique Food Matrix on Human Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB2018-0755D
Record Dates: First submitted 2021-03-09; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Cholesterol, LDL; Cholesterol, HDL; Research Subjects

STUDY DESIGN:
Intervention Model Description: The study design is a two-period, randomized crossover design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant identities were coded and treatments were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-fat ground beef (Experimental): Participants will consume 25 low-fat ground beef patties, 5 patties per week for 5 weeks.
  Interventions: Dietary Supplement: Low-fat ground beef
- High-fat ground beef (Experimental): Participants will consume 25 high-fat ground beef patties, 5 patties per week for 5 weeks.
  Interventions: Dietary Supplement: High-fat ground beef

INTERVENTIONS:
Dietary Supplement: Low-fat ground beef — 5% fat ground beef
  Arms: Low-fat ground beef
Dietary Supplement: High-fat ground beef — 25% fat ground beef
  Arms: High-fat ground beef

SUMMARY:
The primary goal of the proposed research is to document changes in plasma lipoprotein fractions, including high-density lipoprotein (HDL) and low-density lipoprotein (LDL) particle sizes and functionality, following the ground beef interventions. This specifically addresses the hypothesis that increasing the amount of fat in ground beef reduces risk factors for cardiovascular disease. Also, the investigators will measure changes in glucose, insulin, and triacylglycerols (TAG) following low-fat and high-fat ground beef interventions. An important aspect of this research is that the investigators will confirm that consumption of high-fat ground beef will reduce carbohydrate intake and increase insulin sensitivity in men. Furthermore, the investigators will be able to establish which protein sources are voluntarily replaced by the low- and high-fat ground beefs.

DETAILED DESCRIPTION:
Healthy, non-smoking males will be screened for eligibility, and a minimum of 30 males will be selected for the study based primarily on plasma low-density lipoprotein cholesterol (LDL-C) concentrations but also on plasma TAG concentrations. The men must not be consuming restrictive diets or cholesterol-lowering medications, and must not have total cholesterol above 300 mg/dL or below 120 mg/dL. Participants will be requested not to change their habitual level of physical activity. Plasma TAG should not exceed 220 mg/dL. A two-period, randomized cross-over design will be used based on previous studies from our laboratory. Each participant will complete two, 5-week ground beef interventions in a randomly assigned order with a 4-week washout period between the test periods. The men will consume 5 ground beef patties per week for 5 weeks for each ground beef type (25 patties for each type). The two treatments will be low-fat (5% fat) and high-fat (25% fat) ground beef. Participants will be assigned to one of two groups (n ≥ 15 per group), which will be balanced with regard to LDL-C concentrations at the initial screening. The groups will be blocked for age and body weight.

Visit 1 for the subjects selected for the study (immediately before the first dietary intervention) (about 1 hour):

The Registered Dietitian will provide diet instructions, sample menus and cooking instructions. Participants will receive instructions for completion of the diet records using the NutriBase software.

Participants will receive the first set of patties. Subjects will complete a 3-day diet record in NutriBase (which is done at home) before they begin eating the patties. Instructions will also be provided to subjects regarding schedule of patty consumption.

Subjects will complete a 3-day diet record in NutriBase during week 5 of the patty consumption.

The Registered Dietitian or Principal Investigator will contact the study subjects (phone or email) once weekly to ask if the subjects have any questions about the study or the NutriBase system, and ensure they are cooking and using the patties as instructed.

After the initial 5 week intervention, there is a 4 week washout period where subjects will have no study visits and will eat their regular diet. Subjects will be asked to continue complete a 3-day diet record in NutriBase during the last week of the washout period.

The Registered Dietitian or PI will contact the study subjects (phone or email) once weekly to ask if the subjects have any questions about the study or the NutriBase system, and ensure the subjects are cooking and using the patties as instructed.

Source of ground beef. The source of raw materials for production of the 5 and 25% fat patties will be flank and plate primals from feedlot-fed cattle processed through the Rosenthal Meat Science and Technology Center, Texas A&M University. Primals will be selected from grain-fed cattle finished under typical feedlot condition, fed at the Texas A&M University O.D. Butler Animal Science Teaching and Research Center. Prior to the initiation of each phase of the ground beef interventions, each participant will receive an unlabeled box containing 25 frozen, vacuum packaged patties.

Participants will be trained extensively in the preparation and consumption of the ground beef patties. The Registered Dietitian is an individual consultant who will provide professional input regarding cooking methods and diet record keeping to the subjects. The investigators predict that, under conditions in which energy intake remains constant, the percent energy from fat consumed by the participants will increase while the percent energy from carbohydrates will decrease.

Dietary guidelines and diet records. All participants will receive instructions from an Registered Dietitian for the preparation and consumption of the ground beef, including recipes; the Registered Dietitian also will contact the participants as indicated in the study visits above. Other than the patty consumption, subjects will be told to eat their regular diet. Previous studies of the investigators indicated strong compliance to consumption of the ground beef patties, and indicated no changes to the habitual diets of the participants other than a reduction in the percent of calories from carbohydrates.

For the screening visit, participants will be required to visit the Department of Animal Science for a detailed overview of study, including the goals and anticipated outcomes and collect the vital measurements and blood to determine eligibility.

For visit 1, The study staff will explain the Nutribase software and give detailed instructions for the diet records. The Registered Dietitian will provide instruction and suggestions for recipes, and will emphasize the importance of consuming the test ground at the prescribed intervals. During the course of the two, 5-week test periods, the Registered Dietitian or PI will contact the participants at weekly intervals to answer any questions about the completion of the diet records or beef preparation.

Participants will be asked to complete a 3-day diet record during the week before the diet interventions and during the last week of each intervention to establish nutrient intakes and encourage compliance. The NutriBase software is relatively simple to use and will allow more accurate information about dietary intakes. Daily intake of protein, carbohydrates, and fat will be analyzed using commercial NutriBase software. Diet software used in the previous studies of the investigators provided information about lean, medium-fat, and high-fat meat consumption, but did not allow the investigators to determine which meat sources were being replaced by the test ground beef patties; replacement of customary meat sources (e.g., fish, pork, or poultry) by the test patties will be documented in the current study. Additionally, dietary exchanges (meats, breads, fruit, vegetables, etc.) will be analyzed to document the predicted reduction in carbohydrate intake during the consumption of the test patties.

General blood sampling and analyses. On the days of blood sampling, subjects will be asked to report to the laboratory after an overnight fast (at least 10 hours) restricted to water only. Blood (10 mL) will be collected after 5 minutes of seated rest via venipuncture from the antecubital fossa region into serum separator vacutainer tubes using standard, sterile phlebotomy procedures. Blood samples will be drawn during the screening visit and at visits 2, 3, and 4. A total of approximately 40 mL blood will be drawn from each participant over approximately 15 weeks.

After collection, blood will be allowed to clot at room temperature for 2 hours or chilled at 4°C for serum and plasma separation, respectively, prior to centrifugation in a refrigerated centrifuge for 20 minutes (2,000 × g). One serum separator vacutainer will be transported the same day to a commercial, Clinical Laboratory Improvement Amendments (CLIA) certified laboratory for determination of total cholesterol, HDL-C, LDL-C, and TAG using standard clinical chemistry analyses. Aliquots of serum and plasma from additional vacutainers will be transferred into separate 2-mL freezer vials.

Lipoprotein particle number determination. Lipoprotein particle mass area under the curve will be determined with a continuous gradient generated by analytical ultracentrifugation. This procedure allows for the determination at their specific densities of the total number of particles of very low-density lipoprotein (VLDL), LDL, dense LDL-III, dense LDL-V, HDL, buoyant HDL-2b, and remnant lipoprotein (RLP). The concentrations of LDL-I plus LDL-II can be calculated by difference.

Statistical analyses. Because all subjects will be rotated through both ground beef interventions, the data will be analyzed by a split plot design, with diet as the whole plot and time (habitual diet vs test diet) as the split plot. Power calculations were conducted to estimate the required sample size on the basis of data from our previous studies in which HDL-C was increased 2.8 mg/dL by consumption of 24% fat ground beef compared to habitual diets. Analyses used the following assumptions: power was set at 0.8, and a was set at 0.05. It was estimated that a sample size of 16 was sufficient to test the hypothesis that high-fat ground beef would increase HDL-C concentrations.

ELIGIBILITY:
Inclusion Criteria:

* The participants will be male and not have had total cholesterol above 300 mg/dL or below 120 mg/dL.

Exclusion Criteria:

* The participants will be male and must not have been consuming restrictive diets or cholesterol-lowering medications.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Lipoprotein cholesterol | 10 weeks
  Lipoprotein cholesterol concentrations and density distributions

SECONDARY OUTCOMES:
Dietary intake | 10 weeks
  Percent energy from protein, carbohydrate, and fat
Body mass index | 10 weeks
  Body weight in kilograms and height in meters will be measured to calculate body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B. Smith, Ph.D., Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be shared with the funding agency.

REFERENCES:
- [Result] Gilmore LA, Walzem RL, Crouse SF, Smith DR, Adams TH, Vaidyanathan V, Cao X, Smith SB. Consumption of high-oleic acid ground beef increases HDL-cholesterol concentration but both high- and low-oleic acid ground beef decrease HDL particle diameter in normocholesterolemic men. J Nutr. 2011 Jun;141(6):1188-94. doi: 10.3945/jn.110.136085. Epub 2011 Apr 27. PMID 21525253